CLINICAL TRIAL: NCT06921109
Title: Assessment of the Effectiveness of Virtual Reality as a Learning Tool for Relaxation Techniques in Reducing Pediatric Migraines and Tension Type Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, MICHAUX Romane, PhD Student, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE7072024000055
Record Dates: First submitted 2025-01-17; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Headache; Migraine; Tension Type Headache
Keywords: Virtual Reality
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Relaxation training with VR (Experimental): Psychoeducation sessions Relaxation training using biofeedback and Virtual Reality
  Interventions: Behavioral: Experimental: Relaxation training with VR
- Relaxation training without VR (Active Comparator): Psychoeducation sessions Relaxation training using biofeedback
  Interventions: Behavioral: Experimental: Relaxation training without VR
- Control group (Active Comparator): Psychoeducation sessions
  Interventions: Behavioral: No Intervention: Control group

INTERVENTIONS:
Behavioral: Experimental: Relaxation training with VR — This group will benefit from 8 psychoeducation sessions delivered through video modules viewed alongside the psychologist. In addition, an intervention will be implemented to train the children in abdominal breathing and muscle relaxation. This training will be conducted using biofeedback equipment integrated into various virtual environments. Homework exercises will be assigned to them after each session.
  Arms: Relaxation training with VR
Behavioral: Experimental: Relaxation training without VR — This group will benefit from 8 psychoeducation sessions delivered through video modules viewed alongside the psychologist. In addition, an intervention will be implemented to train the children in abdominal breathing and muscle relaxation. This training will be conducted using biofeedback equipment displayed on a computer screen. Homework exercises will be assigned to them after each session.
  Arms: Relaxation training without VR
Behavioral: No Intervention: Control group — This group will benefit from 8 psychoeducation sessions delivered through video modules sent to their homes.
  Arms: Control group

SUMMARY:
The goal of this interventional study is to assess the efficacy of a therapeutic intervention aimed at diminishing pediatric chronic headache. This intervention is based on the development of relaxation skills, particularly the practice of deep breathing, using virtual reality in conjunction with a biofeedback device. Specifically, it aims to assess the relevance of this tool both in learning relaxation techniques and in changing cognitions involved in pain adjustment, such as self-efficacy and pain catastrophizing.

The main hypothesis is that the intervention using virtual reality will lead to greater daily use of the relaxation techniques learned, as well as an increase in the associated self-efficacy, resulting in a reduction in headaches (in terms of frequency and intensity) both immediately after the intervention and two months later.

A secondary hypothesis is that this intervention will contribute to a decrease in negative pain perceptions, pain catastrophizing, and functional disability.

A tertiary hypothesis is that the intervention will lead to an improvement in the child's quality of life.

The effects of this intervention will be compared to those of a similar intervention without the use of virtual reality, as well as to a control condition in which only psychoeducation is provided.

ELIGIBILITY:
Inclusion Criteria:

* Having a history of headaches for at least 6 months, or having been diagnosed with migraines and/or chronic tension-type headaches according to the criteria of the International Headache Society (IHS) by a pediatric neurologist.

Exclusion Criteria:

* having an epilepsy disorder

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of headaches | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  The frequency of headaches is assessed using a sociodemographic questionnaire.
Intensity of headaches | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  The intensity of headaches is assessed using a sociodemographic questionnaire, measured on a Visual Analogue Scale (VAS) ranging from 0 to 10.
Self-efficacy | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  The child's self-efficacy related to functioning while in pain is measured using the Pediatric Rating of Chronic Illness Self-Efficacy (PRCISE). This self-report tool consists of 15 items rated on a Likert-type scale ranging from 0 ("Not at all sure") to 10 ("Very sure"). Higher scores indicate greater self-efficacy.
Coping strategies for pain management | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  The coping strategies used for pain management are assessed using the KidCope questionnaire. This questionnaire evaluates the coping strategies used to address major health concerns that have affected the child over the past month (distraction, social withdrawal, cognitive restructuring, self-criticism, blaming others, problem solving, emotional regulation, wishful thinking, social support, and resignation).
  There exists two versions of the questionnaire. The first is designed for children aged 7 to 12 years and consists of 15 items. The second is tailored for adolescents aged 13 to 18 years and includes 10 items. In both versions, participants indicate whether they use each strategy and whether it helps them manage their pain.
  Scores are calculated for three subscales: positive coping, avoidant coping and negative coping. A higher score indicates a greater tendency to use the assessed coping approach.
Daily diary | During the 8-week intervention (for all three groups) and during the 2 months following the intervention (only for the intervention groups).
  A daily diary assessing the occurence of headaches (frequency and intensity) and the use of coping strategies (frequency and perceived usefulness). This requires the child to document their experiences on a daily basis.
Intervention satisfaction | T1 (Right after the 8-weeks intervention for the experimental groups)
  A customized satisfaction questionnaire regarding the intervention.
Sense of presence questionnaire | 5 minutes after the use of virtual reality during each of the 8 sessions of the virtual reality interventional group
  This questionnaire assesses the sense of presence experienced during the VR immersion. It consists of 16 items, each rated on a Likert-type scale ranging from 0 ("Strongly disagree") to 4 ("Strongly agree"). Scores range from 0 to 64, with higher scores indicating a stronger sense of presence.
Change in simulator sickness questionnaire | Before and 5 minutes after the use of virtual reality during each of the 8 sessions of the virtual reality interventional group
  Change in simulator sickness using the Simulator Sickness Questionnaire (SSQ) which is an instrument used to measure the extent to which children feel simulator sickness due to their immersion in VR (e.g., nausea, eye fatigue, dizziness, etc.). This questionnaire consists of 10 items rated on a Likert-type scale from 0 ("No") to 2 ("A lot"). Scores range from 0 to 20, with higher scores indicating a greater presence of simulator sickness symptoms.

SECONDARY OUTCOMES:
Pain representations | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  Children's pain perception is assessed using the Pain Perceptions Questionnaire for Young People (PPQ-YP). This questionnaire includes four sections: Cognitive representation, which evaluates beliefs regarding the consequences of pain, perceived control, illness coherence, and recurrence (scores range from 0 to 100); Emotional representation, which assesses both responsive and anticipatory emotions related to pain, with scores ranging from 0 to 100 for frequency and intensity; Identity, which measures the frequency of symptoms associated with the pain condition and its treatment (scores range from 0 to 15); and Perceived causes of pain.
  Higher scores on the subscales of consequences, illness coherence, and recurrence reflect stronger beliefs about the negative impact of the pain condition, a clearer understanding of the condition, and the perception of a cyclical and recurrent nature. Conversely, higher scores on the control dimension indicate a greater sense of perceived control.
Pain catastrophization | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  Pain catastrophization is measured using the Pain Catastrophizing Scale for Children (PSC-C), which evaluates various thoughts and emotions children may have when experiencing pain. The scale consists of three subscales: rumination, amplification, and helplessness. It includes 13 items rated on a 5-point Likert-type scale. Total scores range from 0 to 52, with higher scores indicating greater levels of pain catastrophizing.
Functional disability | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  Functional disability is assessed using the Child Activity Limitation Interview (CALI-21), a 21-item instrument with 5-point Likert scales. Total scores range from 0 to 52, with higher scores indicating greater limitations.

OTHER OUTCOMES:
Quality of Life | T0 (Before the intervention), T1 (Right after the 8-weeks intervention), and T2 (2 months post-intervention for interventional groups only)
  The quality of life is assessed using the "Inventaire Systémique de Qualité de Vie pour Enfants" (ISQVE). This scale evaluates the quality of life of children across 20 different life domains: sleep, diet, physical pain, health, clothing, physical appearance, bedroom, relationships with grandparents, relationship with mother, relationship with father, relationships with siblings, contact with friends, how my friends talk about me, school, academic performance, sports or physical activities practiced, non-sport extracurricular activities, autonomy, obedience to authority, tolerance to frustration.
  The scale measures where the child perceives themselves, where they set their objective, and the gap between these two.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Sart Tilman, Liege, Belgium